CLINICAL TRIAL: NCT00725244
Title: A Randomized Prospective Study of Endoscopy Bipolar Eletrocoagulation and Argon Plasma Coagulation of Chronic Rectal Bleeding From Radiation Telangiectasias
Brief Title: Trial of Endoscopy Bipolar and Argon of Chronic Rectal Bleeding From Radiation Telangiectasias
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Luciano Henrique Lenz Tolentino, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 556/05
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-07

CONDITIONS: Radiation Injuries; Telangiectasis
Keywords: Radiation Injuries; Telangiectasis; Bipolar Eletrocoagulation; Argon Plasma Coagulation
MeSH Terms: conditions — Radiation Injuries; Telangiectasis | interventions — Argon Plasma Coagulation; Lasers, Gas

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Bipolar Eletrocoagulation was performed with a high-frequency electrosurgical generator (ERBE® ICC 200 Eletromedizin, Tubingen, Germany), using Gold probe (Wilson- Cook®) with 7 Fr diameter and 300 cm length. The power setting was 50 W. Coagulation of each telangiectasia was achieved with the probes by applying light pressure directly on the telangiectasia.
  Interventions: Device: Bipolar eletrocoagulation
- 2 (Active Comparator): Argon Plasma Coagulation was delivered using a "spray-painting" technique, with short applications at 40 W power with a gas flow of 1.0l per minute. APC equipment was an argon delivery unit (ERBE® ICC 300) coupled a high frequency surgery unit (ERBE® ICC 200). Only the end-firing probe with 2.3 mm and 220 cm length was used. The probe was purged with argon, tested and passed though the endoscope until it extends approximately 1 cm from the tip. The probe was hold just above the mucosal surface and the contact was avoided. During the procedure periodic suction was made to prevent over-distention with gas and consequently patient discomfort.
  Interventions: Device: Argon Plasma Coagulation

INTERVENTIONS:
Device: Bipolar eletrocoagulation — Bipolar Eletrocoagulation was performed with a high-frequency electrosurgical generator (ERBE® ICC 200 Eletromedizin, Tubingen, Germany), using Gold probe (Wilson- Cook®) with 7 Fr diameter and 300 cm length. The power setting was 50 W. Coagulation of each telangiectasia was achieved with the probes by applying light pressure directly on the telangiectasia.
  Other Names: - bipolar probe; - bipolar electrocoagulation
  Arms: 1
Device: Argon Plasma Coagulation — Argon plasma coagulation was delivered using a "spray-painting" technique, with short applications at 40 W power with a gas flow of 1.0l per minute. APC equipment was an argon delivery unit (ERBE® ICC 300) coupled a high frequency surgery unit (ERBE® ICC 200). Only the end-firing probe with 2.3 mm and 220 cm length was used. The probe was purged with argon, tested and passed though the endoscope until it extends approximately 1 cm from the tip. The probe was hold just above the mucosal surface and the contact was avoided. During the procedure periodic suction was made to prevent over-distention with gas and consequently patient discomfort.
  Other Names: Argon Laser; Argonio
  Arms: 2

SUMMARY:
Aim:

To compare the efficacy, safety and number of sessions of bipolar eletrocoagulation (BEC) and argon plasma coagulation (APC) in the management of the bleeding telangiectasias from chronic radiation coloproctopathy (CRCP).

Methods:

Thirty patients with active bleeding from telangiectasias were enrolled in two groups (15 BEC and 15 APC) and classified according of Saunders score. BEC settings were 50 W and APC settings were 40 W and 1.0 l/min. Colonoscopy was the first exam to rule out synchronous lesions and follow-up was performed with sigmoidoscopies. Clinical cure was defined as cessation of bleeding and endoscopic cure was determined by absence of telangiectasias. Failure was defined whenever more than 7 sessions or other therapy was necessary.

DETAILED DESCRIPTION:
Thirty patients with active and chronic hematochezia from radiation telangiectasias were randomized in two groups :

* fifteen patients in group 1- bipolar eletrocoagulation (BE) and
* fifteen in group 2 - argon plasma coagulation(APC). For inclusion in the study, all patients were required to have active (at least one episode last week) and chronic (persist or appear 6 months after the conclusion of radiotherapy) rectal bleeding. Between May 2005 and April 2008, patients were treated and followed at the Endoscopy Unit in the São Paulo Hospital (UNIFESP).

ELIGIBILITY:
Inclusion Criteria:

* active (at least one episode last week) and chronic (persist or appear 6 months after the conclusion of radiotherapy) rectal bleeding.
* previous radiotherapy at least 6 months ago
* presence of colonic or rectal telangiectasias
* patients that agreed to participate of the study and signed the Term of Free Consent and Cleared

Exclusion Criteria:

* prior endoscopic treatment
* rectal or colonic surgery
* stenosis rectal
* rectal bleeding before radiotherapy
* severe cardiac disease

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-05; Primary Completion 2007-11 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Improve of rectal bleeding | 6 months

SECONDARY OUTCOMES:
Complications of each group | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Ferrari, PhD, Study Director — Federal University of São Paulo
Locations (1):
- Federal University Of São Paulo - Gastroenterology, São Paulo, São Paulo, Brazil